CLINICAL TRIAL: NCT00995462
Title: Prevention of Weight Gain in University Students
Acronym: PGP2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marie-France Hivert (Other)
Collaborators: Canadian Diabetes Association (Other); Danone Institute (Unknown)
Responsible Party: Sponsor-Investigator, Marie-France Hivert, MD, Université de Sherbrooke
Organization: Université de Sherbrooke (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 05-025
Record Dates: First submitted 2009-10-14; First posted 2009-10-15 (Estimated); Last update posted 2013-12-11 (Estimated); Status verified 2013-12

CONDITIONS: Prevention; Weight Gain
MeSH Terms: conditions — Weight Gain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (No Intervention)
- Small-group seminar for 2 years (Experimental)
  Interventions: Behavioral: Lifestyle intervention seminars
- Small-group seminars for 1 year followed by email intervention (Experimental)
  Interventions: Behavioral: Lifestyle intervention seminars

INTERVENTIONS:
Behavioral: Lifestyle intervention seminars — The first sessions emphasize acquisition of new knowledge during interactive group seminars designed to maximize attendant's participation by adapting wellknown quiz-show or parlour games to deliver key concepts. A number of sessions are aimed at increasing self-efficacy through problem-solving, time-management strategies, individual self monitoring and goal-setting.During the second year, the intervention focuses on maintenance of healthy behaviour with empowerment of the participants using problem-solving, goal-setting, planning, and self-monitoring skills.
  Arms: Small-group seminar for 2 years; Small-group seminars for 1 year followed by email intervention

SUMMARY:
This study assess whether a small-group seminar intervention to prevent weight gain is effective in a general university student population, and to address the relative role of biological vs. lifestyle factors in predicting weight gain in humans.

ELIGIBILITY:
Inclusion Criteria:

* First year students at the Université de Sherbrooke.

Exclusion Criteria:

* Presence of diseases or medications that would be expected to affect weight (cystic fibrosis, diabetes, inflammatory bowel diseases, anorexia nervosa, bulimia, etc.).
* Pregnancy or planning a pregnancy in the next two years.
* Unable to give an informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 319 (Actual)
Dates: Start 2006-09; Primary Completion 2011-10 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Weight change | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Marie-France Langlois, MD, Principal Investigator — Université de Sherbrooke
Locations (1):
- Université de Sherbrooke, Sherbrooke, Quebec, Canada

REFERENCES:
- [Derived] Langlois F, Langlois MF, Carpentier AC, Brown C, Lemieux S, Hivert MF. Ghrelin levels are associated with hunger as measured by the Three-Factor Eating Questionnaire in healthy young adults. Physiol Behav. 2011 Sep 1;104(3):373-7. doi: 10.1016/j.physbeh.2011.04.013. Epub 2011 Apr 22. PMID 21536060